CLINICAL TRIAL: NCT01547494
Title: A Nutritional Intervention for Migraines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physicians Committee for Responsible Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: WCCR-MIG1
Record Dates: First submitted 2012-02-27; First posted 2012-03-07 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Migraines
Keywords: Migraines; Diet, Vegetarian; Diet, Fat-Restricted; Pain
MeSH Terms: conditions — Migraine Disorders; Pain | interventions — Diet, Vegan; Vitamins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dietary Supplement (Placebo Comparator)
  Interventions: Other: Vegan Diet
- Vegan Diet (Experimental)
  Interventions: Dietary Supplement: mixture of omega3 and vitamins

INTERVENTIONS:
Other: Vegan Diet — Vegan diet, which is devoid of animal products and minimal in fat
  Arms: Dietary Supplement
Dietary Supplement: mixture of omega3 and vitamins — mixture of omega3 and vitamins
  Arms: Vegan Diet

SUMMARY:
The purpose of the study is to assess whether, in individuals with migraines, a low-fat, vegan diet improves pain more effectively than a control supplement or a placebo. The principal measures are pain as measured by Visual Analog Scale (VAS) and the change in migraines frequency. The study duration is 36 weeks.

DETAILED DESCRIPTION:
Preliminary evidence suggests that low-fat, vegetarian diets and certain nutritional supplements can help reduce pain and also reduce the need for pain medications for some people. We will ask about 100 people to participate. All of them will get a low-fat, vegan diet and a nutritional supplement (mixture of omega-3 oils and vitamin E or a placebo), although some will get the diet first, and others will get the supplement first. This order in which they will get the diet and the supplement will be determined randomly, that is, by chance (like the toss of a coin). The principal measures are pain as measured by Visual Analog Scale (VAS)and the change in migraines frequency.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of migraine, as defined by the criteria of the second edition of the International Classification of Headache Disorders18

   * At least 5 attacks fulfilling criteria the criteria below
   * Headache attacks lasting 4-72 hours (untreated or unsuccessfully treated)
   * Headache has at least two of the following characteristics:

     * unilateral location
     * pulsating quality
     * moderate or severe pain intensity
     * aggravation by or causing avoidance of routine physical activity (eg, walking or climbing stairs)
   * During headache at least one of the following:

     * nausea and/or vomiting
     * photophobia and phonophobia
   * Not attributed to another disorder
2. Migraines occurring at least twice per month, on average.
3. Age at least 18 years
4. Ability and willingness to participate in all components of the study
5. Willingness to be assigned to either the diet group or supplement group
6. Migraine medications unchanged within last 6 weeks.

Exclusion Criteria:

1. < 18 years of age
2. Alcohol consumption of more than 2 drinks per day or the equivalent, episodic increased drinking (e.g., more than 2 drinks per day on weekends), or a history of alcohol abuse or dependency followed by any current use
3. Use of recreational drugs in the past 6 months (past drug use, if fully recovered, is not a criteria for exclusion)
4. Pregnancy
5. Unstable medical or psychiatric illness
6. Likely to be disruptive in group sessions (as determined by research staff)
7. Already following a low-fat, vegan diet
8. Lack of English fluency
9. Inability to maintain current medication regimen
10. Inability or unwillingness to participate in all components of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Migraines Pain Change in Migraines frequency | Baseline and 4 months
  Pain as measured by VAS score
Change in Migraines frequency | Baseline and 4 months
  the reduction in the number of migraine attacks.

SECONDARY OUTCOMES:
Quality of life | Baseline and 4 months
  Health related quality of life as measured by a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Physicians Committee for Responsible Medicine, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Bunner AE, Agarwal U, Gonzales JF, Valente F, Barnard ND. Nutrition intervention for migraine: a randomized crossover trial. J Headache Pain. 2014 Oct 23;15(1):69. doi: 10.1186/1129-2377-15-69. PMID 25339342